CLINICAL TRIAL: NCT06771687
Title: High Intensity Interval Training in Patients With a Right Ventricle to Pulmonary Artery Conduit
Acronym: Right HIIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Beatrijs Bartelds, Principal investigator, pediatric cardiologist, associate professor, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MEC-2023-0777
Record Dates: First submitted 2024-09-16; First posted 2025-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease; Truncus Arteriosus; Pulmonary Atresia; Tetralogy of Fallot
Keywords: Heart Defects, Congenital; Truncus Arteriosus, Persistent; Pulmonary Atresia; Tetralogy of Fallot; Physical Conditioning, Human; High-Intensity Interval Training; Exercise Test
MeSH Terms: conditions — Heart Defects, Congenital; Truncus Arteriosus, Persistent; Pulmonary Atresia; Tetralogy of Fallot; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into the intervention or control arm. After the control period, participants in the control arm will also receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm receives the 12-week exercise intervention, with a study visit before and after the intervention.
  Interventions: Behavioral: High intensity interval training
- Control (No Intervention): This arm starts with a 12-week control period, after which the participants will also receive the 12-week exercise intervention. Participants will have a study visit before and after the control period and after the intervention. For the primary outcome parameter, only the control period will be used to compare to the intervention. For the secondary outcome parameters (predictors for response), also the intervention period of the control group will be used.

INTERVENTIONS:
Behavioral: High intensity interval training — A 12-week high intensity interval training program, with 30 minutes of exercise three times a week. The trainings can be completed at home and will be digitally supervised.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if a specific type of exercise training (high intensity interval training) can improve exercise capacity in people with a congenital heart defect that required the creation of a new connection between the right ventricle and pulmonary artery. This includes people with a truncus arteriosus, pulmonary atresia with a ventricular septal defect or severe tetralogy of Fallot. This study focuses on people aged 12 to 45 years. The main questions it aims to answer are:

* Can a 12-week home-based high intensity interval exercise training program increase the exercise capacity?
* Can factors that predict whether or not the exercise training program can increase the exercise capacity in specific people be identified?

Researchers will compare the results from the intervention group to the control group. Participants will be assigned to one of these two groups at inclusion. The control group will also receive the intervention, after the control period.

Participants will:

* Participate in a 12-week home-based exercise training program (3x30 minutes a week, digitally supervised);
* Attend 2 or 3 study visits (which partially is standard care) (2 visits for the intervention group, 3 visits for the control group);
* Each study visit includes: echocardiography, magnetic resonance imaging (MRI) of the heart, cardiopulmonary exercise testing (CPET), blood and feces sampling, and questionnaires on quality of life and physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Congenital absence of an unobstructed connection between the right ventricle and pulmonary artery, requiring surgical implantation of a right ventricle to pulmonary artery conduit, including patients with:

   1. Truncus arteriosus
   2. Pulmonary atresia with ventricular septum defect
   3. Severe tetralogy of Fallot
   4. Other forms of pulmonary atresia with biventricular correction
2. Age 12 to 45 years.
3. Current follow-up in Academic Center for Congenital Heart Disease (ACAHA; Erasmus MC Rotterdam and Radboudumc Nijmegen).
4. Signed informed consent.

Exclusion Criteria:

1. Ventricular arrhythmias and/or channelopathy.
2. Implantable cardioverter defibrillator implantation due to inherited arrhythmia syndromes.
3. Left ventricular ejection fraction and/or right ventricular ejection fraction less than 30 percent.
4. Elite athletes (i.e. national team, Olympians, professional athletes, exercising equal to or more than 10 h/week, according to definition in 2020 European Society of Cardiology Guidelines for Sports Cardiology and Exercise in Patients with Cardiovascular Disease).
5. Cardiovascular lesions requiring intervention (according to international guidelines).
6. Cardiovascular intervention (surgery or catheterization) less than 6 months ago.
7. Cardiovascular medication changes less than 3 months ago.
8. Hospitalization for treatment of cardiovascular events less than 6 months ago.
9. Comorbidities or developmental delay impeding exercise training (e.g. neuromuscular disease, symptomatic myocardial ischemia, syndromic diagnoses such as trisomy 21).
10. Inability to provide informed consent.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption | At baseline, week 14, week 27 (control arm only) and 1 year
  Peak oxygen consumption obtained with CPET

SECONDARY OUTCOMES:
Maximum wattage | At baseline, week 14, week 27 (control arm only) and 1 year
  Maximum wattage obtained with CPET
Heart rate recovery | At baseline, week 14, week 27 (control arm only) and 1 year
  Heart rate recovery obtained with CPET
Ventilatory efficiency slope | At baseline, week 14, week 27 (control arm only) and 1 year
  Ventilatory efficiency slope obtained with CPET
Atrial volumes | At baseline, week 14, week 27 (control arm only) and 1 year
  Atrial volumes obtained with echocardiography
Left and right ventricular inflow pattern | At baseline, week 14, week 27 (control arm only) and 1 year
  Left and right ventricular inflow pattern obtained with echocardiography (E and A waves)
Ventricular size | At baseline, week 14, week 27 (control arm only) and 1 year
  Ventricular size obtained with echocardiography
Left and right ventricular ejection fraction | At baseline, week 14, week 27 (control arm only) and 1 year
  Left ventricular ejection fraction obtained with echocardiography
Right ventricular fractional area change | At baseline, week 14, week 27 (control arm only) and 1 year
  Right ventricular fractional area change obtained with echocardiography
Tricuspid annular plane systolic excursion (TAPSE) | At baseline, week 14, week 27 (control arm only) and 1 year
  TAPSE obtained with echocardiography
Ventricular strain | At baseline, week 14, week 27 (control arm only) and 1 year
  Ventricular strain obtained with echocardiography
Vascular flow | At baseline, week 14, week 27 (control arm only) and 1 year
  Vascular flow (aortic valve, RV-PA conduit, mitral and tricuspid valve) obtained with echocardiography
Ventricular size | At baseline, week 14 and week 27 (control arm only)
  Ventricular size obtained with MRI
Right and left ventricular ejection fraction | At baseline, week 14 and week 27 (control arm only)
  Right and left ventricular ejection fraction obtained with MRI
Ventricular mass | At baseline, week 14 and week 27 (control arm only)
  Ventricular mass obtained with MRI
Vascular flow | At baseline, week 14 and week 27 (control arm only)
  Two-dimensional phase-contrast flow in the aorta and main pulmonary artery, obtained with MRI
Ventricular kinetic energy | At baseline, week 14 and week 27 (control arm only)
  Ventricular kinetic energy obtained with four-dimensional flow MRI
NT-proBNP | At baseline, week 14 and week 27 (control arm only)
  NT-proBNP in blood
GDF-15 | At baseline, week 14 and week 27 (control arm only)
  GDF-15 in blood
Soluble ST-2 | At baseline, week 14 and week 27 (control arm only)
  Soluble ST-2 in blood
Galectin-3 | At baseline, week 14 and week 27 (control arm only)
  Galectin-3 in blood
Gut microbiome composition | At baseline, week 14 and week 27 (control arm only)
  Gut microbiome composition analyzed using 16S rRNA sequencing in fecal samples
Changes in weight | At baseline, week 14, week 27 (control arm only) and 1 year
  Changes in weight (kg) and derivatives such as BMI (weight / height^2, reported in kg/m^2)
Time in moderate-to-vigorous and sedentary activity | At baseline, week 14, week 27 (control arm only) and 1 year
  Average time per day and total time (minutes and percentage), measured by accelerometry with the Actigraph waist accelerometer worn for seven days
Time in moderate-to-vigorous and sedentary activity | At baseline, week 14, week 27 (control arm only) and 1 year
  Measured using the Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH) questionnaire
Quality of life (child perspective) | At baseline, week 14, week 27 (control arm only) and 1 year
  Measured by Child Health Questionnaire (CHQ) Child Form (CF) (CHQ-CF45) for participants aged under 18 years, scale 0-100 (100 being the best outcome)
Quality of life (parent perspective) | At baseline, week 14, week 27 (control arm only) and 1 year
  Measured by Child Health Questionnaire (CHQ) Parent Form (PF) (CHQ-PF28) for participants aged under 18 years, scale 0-100 (100 being the best outcome)
Quality of life | At baseline, week 14, week 27 (control arm only) and 1 year
  Measured by the 36-Item Short Form Health Survey (SF-36) questionnaire for participants aged over 18 years, scale 0-100 (100 being the best outcome)
Fatigue-related quality of life | At baseline, week 14, week 27 (control arm only) and 1 year
  Measured by the PedsQL Multidimensional Fatigue Scale for all participants, scale 0-100 (100 being the best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrijs Bartelds, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - ErasmusMC, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No